CLINICAL TRIAL: NCT00240032
Title: A Double-Blind, Randomized, Placebo Controlled Study of An Oral Antihistamine on Local Injection Site Reactions Among Persons With Multiple Sclerosis Who Perform Daily Injections of Copaxone® Using Autoject® 2 for Glass Syringe.
Brief Title: A Study to Evaluate the Impact on Skin (Injection Site) Reactions of Taking an Antihistamine (Zyrtec®) or Placebo Prior to Daily Injections of Copaxone®.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Thomas Smith, MD, VP Medical Affairs, Teva Neuroscience
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PM014
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Glatiramer Acetate; Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Copaxone® with Zyrtec (Active Comparator)
  Interventions: Drug: glatiramer acetate injection with oral cetirizine hydrochloride
- Copaxone® with placebo (Experimental)
  Interventions: Drug: glatiramer acetate with placebo

INTERVENTIONS:
Drug: glatiramer acetate injection with oral cetirizine hydrochloride — Copaxone® injection 20 mg, Oral Zyrtec® 10 mg tablet
  Other Names: Copaxone®, Zyrtec®
  Arms: Copaxone® with Zyrtec
Drug: glatiramer acetate with placebo — Copaxone® injection 20 mg, oral placebo
  Other Names: Copaxone®
  Arms: Copaxone® with placebo

SUMMARY:
This study is designed to compare injection skin (injection site) reactions when an antihistamine (Zyrtec®) or placebo is taken prior to performing daily Copaxone® injections. Patients will be assigned (like a flip of a coin) to take either a placebo or an antihistamine (Zyrtec®) prior to performing their daily Copaxone® injections. The patient and physician will be unaware whether they are taking a placebo or antihistamine during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 18 years of age or older
* Diagnosis of RRMS
* Beginning or recently (within < 3months) began self-injecting Copaxone®

Exclusion Criteria:

* Taking any other immunomodulatory therapy in conjunction with Copaxone®
* Unable to perform subcutaneous self-injection
* Pregnant or trying to become pregnant, or breast feeding during the study
* Previously participated in this study or in another clinical trial in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-10; Primary Completion 2006-06 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Injection Site Reaction | 5 weeks
  Injection site reaction after taking antihistamine

CONTACTS AND LOCATIONS:
Overall Officials: MerriKay Oleen-Burkey, Ph.D., Study Director — Teva Neuroscience, Inc.